CLINICAL TRIAL: NCT02241941
Title: Evaluation of Single-dose Pharmacokinetics of Intravenous Daptomycin in Patients With Thermal Injury
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Assessment of daptomycin concentrations with microdialysis technically not feasible
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dapto-ICU-09; EK-1748
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Burn Injury
MeSH Terms: conditions — Burns | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daptomycin (Experimental)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin

SUMMARY:
The purpose of this study is to determine single dose pharmacokinetics of daptomycin consecutively in 10 patients on three different time points after severe burn injury.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of 18 years or older
* Second and/or third degree thermal injury
* Total body surface area burned ≥ 15%
* Hospitalisation in the ICU for burn injured patients of the University Hospital Zürich
* Probability of ICU stay of >14 days
* Written informed consent by the patient or in patients unable to be informed or to sign according to section 4.4 of the study protocol

Exclusion Criteria:

* Evidence of renal failure (Creatinine clearance <30ml/min) or continuous renal replacement therapy such as continuous hemofiltration
* History of muscle disease or skeletal muscle disorder
* Creatine-phosphokinase (CPK) ≥ 5 times the upper limit of normal (ULN)
* History of hypersensitivity to the drug
* Pregnancy
* Severe coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of daptomycin | up to 30 days

SECONDARY OUTCOMES:
Correlation of daptomycin plasma concentrations with tissue concentration | up to 30 days
degree of variability of daptomycin pk parameters in dependency of body surface area burned | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Weber, MD Professor, Principal Investigator — Division of Infectious Diseases and Hospital Epidemiology, Universitit Hospital Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland